CLINICAL TRIAL: NCT00404599
Title: A Randomised, Double Blind, Parallel-Group Study of the Oxidative Stress Lowering Effect of Simvastatin and Atorvastatin.
Brief Title: Oxidative Stress Lowering Effect of Simvastatin and Atorvastatin.
Acronym: SOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Dr. Y . Smulders, Vu University medical centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABR 15330
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: simvastatin, atorvastatin, oxidative stress
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Atorvastatin; Simvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: atrorvastatin 10mg — Atorvastatin 10 mg once a day
  Other Names: Lipitor
Drug: simvastatin 40mg — simvastatin 40mg once a day
  Other Names: Zocor

SUMMARY:
Background: HMG-CoA reductase inhibitors (statins) are effective lipid-lowering agents and are known to reduce cardiovascular events. Beneficial effects of statins seem to occur very early in the course of their therapy and subgroup analysis of large trials indicates that subjects in statin-treated arms have less cardiovascular events than subjects in placebo-controlled arm with comparable serum cholesterol levels. Therefore, it has been suggested that statins may have antiatherogenic effects beyond their cholesterol lowering effect. Many studies have demonstrated a rapid improvement in vascular function with atorvastatine which cannot solely be accounted for by achieved lipid reduction. A rapid oxidative stress lowering effect of atorvastatin has been proposed as the probable mechanism of this action. Whether atorvastatine has stronger antioxidant effect and whether atorvastatin lowers oxidative stress earlier in the course of therapy than other statins has not been studied yet.

Objective: To compare the rapidity of onset and the extent of oxidative stress lowering of atorvastatin with that of an (in terms of LDL lowering) equipotent dosage of simvastatin.

Methods: We plan to recruit sixty statin naive patients, with diabetes mellitus type 2 and/or obesity (BMI > 25) and/or hypertension (RR>140/90 mmHg). Patients with K/DOQI stage 5 chronic kidney disease (Cockcroft-Gault clearance of less than 15 ml/min/1.73m2), patients who use any vitamin preparation, or statins in the last three months and patients with LDL cholestrerol < 2.5 mmol/l will be excluded from the study. Because of the influence of angiotensin-converting enzyme inhibitors (ACE-inhibitors) on oxidative stress, patients will be stratified for prior ACE-inhibitor use during randomization. All included patients are randomized to treatment with simvastatin 40 mg daily or atorvastatin 10 mg daily to achieve a comparable lipid reduction. Established parameters of oxidative stress such as oxidized LDL, malondealdehyde and isoprostane will be measured in plasma on inclusion, one week, six weeks and three months after inclusion. We also plan to measure endothelial function parameters such as soluble Vascular Adhesion Molecule (sVCAM) and von Willebrand factor. In addition, parameters of inflammation such as high sensitive C - reactive protein, TNF-alfa, interleukin-6 and myeloperoxidase will be measured to investigate whether there is any correlation between oxidative stress lowering and endothelial function and inflammation. The inhibitory effect of HDL to prevent oxidation of LDL will be determined by measurement of lipid peroxides formed during in vitro oxidation of LDL co-incubated with HDL. The inflammatory / anti-inflammatory properties of HDL will be tested by measurement of the HDL capacity to inactivate oxidized palmitoyl-2-arachidonoyl-sn-glycero-3-phosphorylcholine (ox-PAPC). Collections of 24 hours of urine at the beginning and after one week, six weeks and three months will be used to measure urine F2-isoprostane levels.

Analyses: All parameters of oxidative stress before and during treatment with both statins will be compared to determine whether atorvastatin causes a stronger and quicker reduction of oxidative stress than simvastatin. Generalized estimating equations (GEE) will be used to compare these effects. We plan to include a minimum of 30 patients in each treatment-group from the outpatient clinic of the department of internal medicine of the VU University Medical Center in Amsterdam.

Expected results: Atorvastatin will reduce oxidative parameters stronger and earlier than simvastatin.

DETAILED DESCRIPTION:
Background HMG-CoA reductase inhibitors (statins) are effective lipid-lowering agents and are known to reduce cardiovascular events. It was initially assumed that cholesterol reduction by statins was the only mechanism responsible for their beneficial effect. However, beneficial effects of statins seem to occur very early in the course of their therapy [1] and subgroup analysis of large trials indicates that subjects in statin-treated arms have less cardiovascular events than subjects in placebo-controlled arm with comparable serum cholesterol levels [2]. Therefore, it was suggested that statins may have antiatherogenic effects, such as anti-inflammatory and antioxidative actions, beyond their cholesterol lowering effect. Many studies have demonstrated a rapid improvement in vascular function with atorvastatine which cannot solely be accounted for by achieved lipid reduction [3-5]. In the Pravastatin or Atorvastatin evaluation and infection therapy-thrombolysis in myocardial infarction 22 trial (PROVE-IT-TIMI 22 trial), with a follow-up period of 2-years and intensive statin therapy, 80 mg atorvastatin showed a stronger reduction of cardiovascular events when compared with 40 mg pravastatin, with an apparent benefit observed early [6]. A rapid and a strong oxidative stress lowering effect of atorvastatin has been proposed as the probable mechanism of this action [7]. Other statins have been shown to have anti-oxidant effects as well [8,9]. However, whether atorvastatine has stronger antioxidant effect and whether atorvastatin lowers oxidative stress early in the course of therapy than other statins has not been demonstrated up to now.

Hypothesis: Atorvastatin shows a more rapid and stronger antioxidative effect compared to simvastatin.

Study objective The objective of this study is to compare the oxidative stress lowering capacity of atorvastatin, the most widely used statin in the US, with that of simvastatin in a population of patients with increased oxidative stress (in patients with diabetes mellitus [10], hypertension [11] obesity [12] and chronic kidney disease [13] who are known to have increased oxidative stress).

Design and methods We plan to recruit sixty statin naive patients with diabetes mellitus type-2 and/or obesity (BMI > 25 kg/m2) and/or hypertension (RR> 140/90 mmHg). Patients with K/DOQI stage 5 chronic kidney disease (Cockcroft-Gault clearance of less than 15ml/min/1.73m2) and patients who use any vitamin preparation or statins in the last three months will be excluded from the study. Because of the documented influence of ACE-inhibitors on oxidative stress we will stratify patients for prior ACE-inhibitor use during randomization. All included patients are randomized to treatment with simvastatin 40 mg daily or atorvastatin 10 mg daily in order to achieve a comparable lipid reduction. Established parameters of oxidative stress, such as oxidized LDL, malondealdehyde will be measured (14-18) in plasma on inclusion, one week, six weeks and three months after the inclusion. Primary end point of the study will be the absolute difference between oxidized LDL reduction between the two groups. We also plan to measure endothelial function parameters such as soluble Vascular Adhesion Molecule (sVCAM) and von Willebrand factor. In addition parameters of inflammation such as high sensitive c-reactive protein, TNF-alfa and Interleuking-6 will also be measured to investigate whether there is any correlation between eventual oxidative stress lowering and endothelial function and inflammation. The inhibitory effect of HDL to prevent oxidation of LDL will be determined by measurement of lipid peroxides formed during in vitro oxidation of LDL co-incubated with HDL. The anti-inflammatory properties of HDL will be tested by measurement of the HDL capacity to inactivate oxidized palmitoyl-2-arachidonoyl-sn-glycero-3-phosphorylcholine (ox-PAPC). For this measurement we will use a cell-free assay that has been developed by Navab and co-workers (19). Collections of 24 hours of urine at the beginning and after one week, and three months will be used to measure urine F2-isoprostane levels (20-24).

Power calculation:

The number of patients needed to detect an absolute Oxidized LDL difference of 9 U/L between the two groups over 3 months with a power of 80%, α of 0.05 and a SD of 12 was 30 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Hypertension

Exclusion Criteria:

* chronic kidney disease K/DOQI stage 5
* use of statins

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in oxLDL levels | july 2009

SECONDARY OUTCOMES:
Reduction in plasma malondialdehydes and urine isoprostanes | july 2009
Reduction in plasma endothelial function parameters such as soluble Vascular Adhesion Molecule (sVCAM) and von Willebrand factor | july 2009

CONTACTS AND LOCATIONS:
Overall Officials: Prabath Nanayakkara, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands